CLINICAL TRIAL: NCT02150577
Title: Partnership for Implementation of Evidence-Based Practices in Rural Primary Care
Brief Title: Implementation Trial of Evidence Based Practices for Mood Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MH085104
Record Dates: First submitted 2014-05-27; First posted 2014-05-30 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Bipolar Disorder; Treatment Resistant Depression
Keywords: Screening; Mood Stabilizers; Computer delivered psychotherapy; Peer Support; Telepsychiatry; Implementation; Rural
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Implementation (Experimental): Evidence Based Quality Improvement
  Interventions: Behavioral: Evidence Based Quality Improvement
- Control (No Intervention): Usual Quality Improvement

INTERVENTIONS:
Behavioral: Evidence Based Quality Improvement — Facilitation of the identification, adoption, adaption and implementation of evidence based practices.
  Arms: Implementation

SUMMARY:
The objective of this Implementation Trial is to evaluate the implementation of evidence based practices for Bipolar Disorder and Treatment Resistant Depression in small rural Federally Qualified Health Centers. The evidence based practices chosen and adapted by Health Center providers and patients in consultation with clinical experts include: screening for and diagnosing Bipolar Disorder, prescribing mood stabilizers, on-line cognitive behavioral therapy, on-line peer support, collaborative care management and tele-psychiatry consultation. A quasi-experimental study design will be used, with each of the six participating Federally Qualified Health Centers choosing one implementation clinic and one control clinic. Implementation outcomes include: reach, adoption, implementation-fidelity and effectiveness. Providers and patients may choose to use all, any or none of the evidence based practices based on their needs and preferences. Data will be collected from chart review and patient surveys will be administered by an Interactive Voice Response telephone system.

DETAILED DESCRIPTION:
The objective of this Implementation Trial is to evaluate the implementation of evidence based practices for Bipolar Disorder and Treatment Resistant Depression in small rural Federally Qualified Health Centers. The evidence based practices were chosen and adapted by Health Center providers and patients in consultation with clinical experts. The evidence based practices include: screening for and diagnosing Bipolar Disorder, prescribing one of five mood stabilizers, on-line cognitive behavioral therapy (Beating the Blues), on-line peer support (Depression and Bipolar Support Alliance), collaborative care management and tele-psychiatry consultation. These evidence based practices were chosen based on the strength of the research evidence and the feasibility of implementation in small primary clinics serving a low income rural patient population. Providers may choose to use all, any or none of the evidence based practices with their patients. Patients may choose to adhere to all, any, or none of the treatment recommendations prescribed by their provider.

A quasi-experimental study design will be used. There are Federally Qualified Health Centers participating in the Implementation Trial. Each Federally Qualified Health Center chose one implementation clinic and one control clinic. Patients will be enrolled from both implementation and control clinics and outcomes will be compared for the three month period following enrollment. Implementation outcomes are based on the "RE-AIM" framework and include: reach, adoption, implementation-fidelity and effectiveness. Reach represents the proportion of patients who receive evidence based practices. Reach will be compiled at the patient level. Adoption represents the proportion of providers delivering evidence based practices. Provider adoption will be compiled at the primary care provider level. Implementation-Fidelity represents whether the evidence based practices are being delivered as intended. Implementation will be compiled at the patient level. Effectiveness represents the clinical improvement experienced by patients. Effectiveness will be compiled at the patient level. Data will be collected from chart review and patient surveys will be administered by an Interactive Voice Response telephone system.

There will be three samples. The Full Sample will be all patients screening positive for depression on the Patient Health Questionnaire (PHQ9) screening tool during the 9 month enrollment period. The PHQ9 is used to routinely screen patients for depression at participating clinics. The Full Sample is expected to include approximately 2,400 patients. The Bipolar Depression Sample will be patients screening positive for depression, screening positive for Bipolar Disorder (on the CIDI), and providing informed consent to collect primary data. The Treatment Resistant Depression Sample will be patients screening positive for depression, screening negative for Bipolar Disorder, currently prescribed an antidepressant, and providing informed consent to collect primary data. The purpose of the "currently prescribed an antidepressant" inclusion criterion is to identify patients who do not respond to treatment. This inclusion criterion will be determined from chart review. We expect approximately 40 patients from each of six Federally Qualified Health Centers (two clinics per system) to be eligible for the Bipolar Depression and Treatment Resistant Depression samples and to provide informed consent. Thus, the combined size of the Bipolar Depression and Treatment Resistant Depression samples is expected to be 240.

Health Center evaluation staff will test differences in patient outcomes at implementation and control sites using ordinary least squares and logistic regression analyses that will control for demographic characteristics. Compared to patients at control sites, we hypothesize that patients with a positive depression screen at implementation sites will be more likely to be screened for Bipolar Disorder than patients at control sites. With automated chart review data for 2,400 patients, we will have 84% power to detect a 5% (e.g., 25% versus 20%) difference in Bipolar Disorder screening rates. Compared to patients at control sites, we hypothesize that patients in the Bipolar Disorder Sample at implementation sites will be more likely to see receive a Bipolar diagnosis, be prescribed a mood stabilizer, engage in on-line cognitive behavioral therapy, engage in on-line peer support, receive collaborative care management, have a tele-psychiatry consultation, experience depression symptom improvement and report greater satisfaction. For the Bipolar Disorder Sample, we plan to enroll approximately 20 patients from each of six Federally Qualified Health Centers (two clinics per system) and expect at least a 75% follow-up rate (n=90), which will give us 79% power to detect a 25% (e.g., 15% versus 40%) difference in Bipolar Disorder specific outcomes (e.g., diagnosed with Bipolar Disorder). Compared to patients at control sites, we hypothesize that patients in the Treatment Resistant Depression Sample at implementation sites will be more likely to have their antidepressant prescription changed, engage in on-line cognitive behavioral therapy, engage in on-line peer support, receive collaborative care management, have a tele-psychiatry consultation, experience depression symptom improvement and report greater satisfaction. For the Treatment Resistant Depression Sample, we plan to enroll approximately 20 patients from each of six Federally Qualified Health Centers (two clinics per system) and expect at least a 75% follow-up rate (n=90), which will give us 79% power to detect a 25% (e.g., 15% versus 40%) difference in Treatment Resistant Depression specific outcomes (e.g., antidepressant prescription changed). For the combined Bipolar Disorder Sample and Treatment Resistant Depression Sample, we plan to enroll approximately 40 patients from each of six Federally Qualified Health Centers (two clinics per system) and expect at least a 75% follow-up rate (n=180), which will give us 87% power to detect a 15% (e.g., 25% versus 40%) difference in trans-diagnostic outcomes (e.g., satisfaction).

ELIGIBILITY:
Inclusion Criteria:

Full sample - screening positive for depression Bipolar Disorder sample - screening positive for depression, screening positive for bipolar disorder, not currently in a manic state Treatment Resistant Depression - screening positive for depression, screening negative for bipolar disorder, currently prescribed an antidepressant by primary care provider

Exclusion Criteria:

Full sample - none Bipolar Disorder sample - currently in a manic state Treatment Resistant Depression - none

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Patient Reach | 3 months
  For patients in the Bipolar Depression Sample and Treatment Resistant Depression Sample, we will measure psychotherapy reach defined as the percentage of patients who report using the on-line cognitive behavioral therapy computer program. We will measure peer support reach defined as the percentage of patients who report using the Depression and Bipolar Support Alliance website chat room. We will measure tele-psychiatry reach as the percentage of patients who report seeing a tele-psychiatrist. For the Bipolar Depression Sample, we will measure diagnostic reach defined as the percentage of patients who are assigned a Bipolar Disorder diagnosis and mood stabilizer reach as the percentage of patients who are prescribed a mood stabilizer. For the Treatment Resistant Depression Sample, we will measure antidepressant prescription change reach as the percentage of patients who are prescribed a different antidepressant than the one prescribed when they screened positive for depression.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Curran, PhD, Principal Investigator — University of Arkansas
Locations (6):
- United States (6):
  - Mainline Health Systems Inc., Eudora, Arkansas
  - Boston Mountain Rural Health Center, Huntsville, Arkansas
  - Lee County Cooperative Clinic, Marianna, Arkansas
  - ARcare, Melbourne, Arkansas
  - Jefferson Comprehensive Care System, Pine Bluff, Arkansas
  - East Arkansas Family Health Center, West Memphis, Arkansas

REFERENCES:
- [Background] Hunt JB, Curran G, Kramer T, Mouden S, Ward-Jones S, Owen R, Fortney J. Partnership for implementation of evidence-based mental health practices in rural federally qualified health centers: theory and methods. Prog Community Health Partnersh. 2012 Fall;6(3):389-98. doi: 10.1353/cpr.2012.0039. PMID 22982852